CLINICAL TRIAL: NCT04092478
Title: ''Compare Abdominal Crunch Positions With Conventional Sitting and Lateral Decubitus Positions in Terms of Interspinous Distance in Adult Patients''
Brief Title: '' Abdominal Crunch Positions With the Others in Terms of Interspinous Distance in Adult Patients ''
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Yasin TİRE, Principal Investigator, Konya Meram State Hospital
Other Study IDs: YTire
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Traditional Sitting Position: We are going to use the Traditional Sitting Position on each patients.
  Interventions: Other: Spinal Anesthesia Position
- Lateral Decubitis Position: We are going to use the Lateral Decubitis Position on each patients.
  Interventions: Other: Spinal Anesthesia Position
- Abdominal Crunch Position: We are going to use the Abdominal Crunch Position on each patients.
  Interventions: Other: Spinal Anesthesia Position

INTERVENTIONS:
Other: Spinal Anesthesia Position — The patient positions during the spinal anesthesia

SUMMARY:
The most important factor for ease of operation and safety during spinal anesthesia is the determination of the spinal space. Increasing lumbar flexion facilitates access to the spinal space. Traditionally, patients undergo spinal anesthesia with lateral or sitting lumbar flexion.

In a study by Martha L Walker et al., The maximum extension of the knees, adduction of the hip, and a modified sitting position with the back flexion, ie, the abdominal crunch position, were found to be effective in increasing the flexion of the lumbar spine.

In our study, we aimed to measure the interspinal distance with the abdominal crunch position with the help of ultrasonography (USG) and to compare the interspinal distance with the measurements obtained in traditional positions (sitting position and lateral decubitus).

DETAILED DESCRIPTION:
Interspinal distance will be measured by ultrasonography by 3 different positions, respectively, for the patients who will undergo elective surgery and meet the study criteria and give voluntary consent.

This evaluation process is to record and compare the measurement results. Patients will not undergo any interventional procedures.

Patients who have difficulty in positioning due to hip, femur, knee and tibial fractures or arthrosis and who cannot be communicated will not be included in the study.

One hundred of patients over the age of 18 who will undergo elective surgery will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Undergo elective surgery

Exclusion Criteria:

* Patients with vertebral anomaly
* Patient with not communicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred of patients over the age of 18 who will undergo elective surgery will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Inter spinal distance | Through study completion, an average of 6 months.
  Increasing of the Inter spinal distance

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Tire, MD, Principal Investigator — Konya Meram State Hospital
Locations (1):
- Yasin Tire, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No